CLINICAL TRIAL: NCT06749470
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Study on the Treatment of Depression with Jieyu Chufan Capsules
Acronym: JOYS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Lingjiang Li, Chief physician, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-10-22-674
Record Dates: First submitted 2024-12-23; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Jieyu Chufan Capsules; TCM; Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, multicenter clinical study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Jieyu Chufan Capsules Strength: 0.4 g/capsule, 3 × 12 capsules/plate/box Administration: 4 capsules, tid, 8 weeks
  Interventions: Drug: Jieyu Chufan Capsules
- Control Group (Placebo Comparator): Jieyu Chufan Capsules Placebo Strength: 0.4 g/capsule, 3 × 12 capsules/plate/box. Administration: 4 capsules, tid; 8 week
  Interventions: Drug: Jieyu Chufan Capsules simulant

INTERVENTIONS:
Drug: Jieyu Chufan Capsules — 4 capsules, tid; 8 weeks
  Arms: Test Group
Drug: Jieyu Chufan Capsules simulant — 4 capsules, tid; 8 weeks
  Arms: Control Group

SUMMARY:
To evaluate the efficacy of Jieyu Chufan Capsules, with placebo as the control, in combination with SSRIs in patients with moderate and severe depression.

To observe the safety of Jieyu Chufan Capsules and its effects in improving the side effects of SSRIs.

DETAILED DESCRIPTION:
Major depressive disorder (MDD), a common affective mental disorder caused by a variety of reasons, is mainly clinically manifested as significant and persistent low mood, loss of interest, retardation of thinking, pessimism, lack of initiative, self-guilt, loss of appetite, sleep disorders, and paranoia, often accompanied by various systemic discomfort that is inconsistent with objective examinations, and in severe cases, suicidal thoughts and behaviors[1]. Although there has never been a name called "depression" in ancient literature of traditional Chinese medicine, it has been long recognized since it is similar to many diseases in Chinese medicine literature (such as "depression syndrome" and "lily disease"). Depression is a common mental disorder that affects about one fifth people in a certain period in their lives.

According to the data disclosed by the WHO, there are more than 350 million people suffering from depression in the world, with an increase of about 18% in the past decade. According to the prevalence report of China Mental Health Survey (CMHS) in 2019[2], for depressive disorders, the lifetime prevalence was 6.8% and the 12-month prevalence was 3.6% in China, among which, for depression, the lifetime prevalence was 3.4%, and the 12-month prevalence was 2.1%. With the acceleration of the pace of modern life, its prevalence is spreading. Moreover, the pandemic of COVID-19 resulted in a 27.6% increase in global cases of major depressive disorder[3]. It is estimated that by 2030, depressive disorders will surpass tumors and cardiovascular and cerebrovascular diseases to become the largest disease burden in the world[4]. For the time being, there are limited treatment measures for depressive disorders, and about 30%-40% of patients have developed to refractory depression due to insensitivity to existing monoamine antidepressants[5]. Monoamine antidepressants have shortcomings such as slow action, residual symptoms, more adverse reactions, and long-term medication, while novel fast-acting antidepressants also have the problems of drug addiction and neurotoxicity[6], so its treatment is facing a new dilemma.

Traditional Chinese medicine has been used for prevention and treatment of various depressive disorders for more than two thousand years, and it costs less and has achieved reliable clinical efficacy and caused less toxic side effects. Traditional Chinese medicine believes that emotional factors, such as anger, sorrow, sadness, and too much thinking, result in liver dysfunction, spleen dysfunction, mental dysfunction, and then multiple viscera dysfunction, and long-term liver depression generates pathogenic fire and fire burns body fluid to produce phlegm, thus forming the critical pathogenesis of depression, i.e., qi stagnation, phlegm condensation, and fire stagnation. The prescription of Jieyu Chufan Capsules, originated from the Classical Prescriptions of Zhang Zhongjing, is prepared by modifying the Pinellia and Magnolia Decoction and the Cape jasmine and Magnolia Decoction. Since 1997, modified Jieyu Chufan Capsules has been used to treat 12,000 outpatient cases, including 445 cases of depression and anxiety. The phase III clinical study of Jieyu Chufan Capsules[7] showed that Jieyu Chufan Capsules effectively improved depression and anxiety and effectively alleviated the physical symptoms of patients with mild to moderate depressive disorders, and the incidence of adverse reactions was comparable to that of placebo and significantly lower than that of fluoxetine.

The prescription of Jieyu Chufan Capsules, originated from the Classical Prescriptions and developed based on clinical application, has significant clinical efficacy in clearing heat and relieving fidgetiness, activating qi and eliminating phlegm. The randomized, double-blind, placebo-controlled, multicenter clinical study will be conducted to further evaluate the efficacy and safety of Jieyu Chufan Capsules in the treatment of symptoms related to moderate to severe depression in a wider population. The reliable evidence-based medical evidence can provide reference for clinical application of the drug.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18-65 years (inclusive);
2. With first-episode or relapsed depression that meets the DSM-5 diagnostic criteria;
3. With a Hamilton's Depression Scale (HAMD-17) score of ≥18 at enrollment;
4. Receiving no antidepressants within 2 weeks (fluoxetine within 6 weeks) prior to enrollment;
5. Willing to sign the informed consent form (ICF).

Exclusion criteria:

1. Meeting the DSM-5 diagnostic criteria for mental disorders other than depression (e.g., patients with schizophrenia spectrum and other psychiatric disorders, bipolar and related disorders, compulsive and related disorders, etc.);
2. With refractory depression (no response to adequate treatment with 2 or more antidepressants) as determined by the investigator or previously diagnosed;
3. At a significant risk of suicide (HAMD-17 Item 3 (suicide) score ≥3) as judged by the investigator, or with a history of suicide attempts in the last year;
4. Receiving non-drug therapies, such as electric convulsive therapy (ECT), repetitive transcranial magnetic stimulation (rTMS), and systematic psychotherapy 10 or more times in the last 6 months;
5. With other serious chronic diseases such as severe thyroid disease, Parkinson's disease, tumor, epilepsy, and severe rheumatism;
6. With clinically significant abnormalities in 12-lead ECG that may affect the safety of the subject, including but not limited to acute myocardial ischemia, myocardial infarction, severe arrhythmia, or significantly prolonged QTc (QTc >450 ms in men and >470 ms in women);
7. With severe hepatic and renal insufficiency, i.e., aspartate transaminase (AST) ≥1.5 × upper limit of normal (ULN) or alanine aminotransferase (ALT) ≥1.5 × ULN, and serum creatinine (Scr) ≥1.5× ULN;
8. Allergic to the investigational drug or its ingredients;
9. In lactation, of childbearing potential, or planning to be pregnant;
10. With alcohol and drug dependence;
11. Participating in another clinical study within 1 month prior to enrollment or for the time being.
12. Not suitable for participation in this study due to potential risks or other factors as considered by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-12-22 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HAMD-17 score from baseline at Week 8. | From enrollment to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Response rate in HAMD-17 at Week 8 relative to baseline | From enrollment to the end of treatment at 8 weeks
Remission rate in HAMD-17 at Week 8 relative to baseline | From enrollment to the end of treatment at 8 weeks
Change in HAMA score from baseline at Week 8 | From enrollment to the end of treatment at 8 weeks
Change in QIDS-SR16 score from baseline at Week 8 | From enrollment to the end of treatment at 8 weeks
Change in GAD-7 score from baseline at Week 8 | From enrollment to the end of treatment at 8 weeks
Change in SHAPS score from baseline at Week 8 | From enrollment to the end of treatment at 8 weeks
Change in SDS score from baseline at Week 8 | From enrollment to the end of treatment at 8 weeks

IPD SHARING:
Plan to Share IPD: No
Considering subject privacy